CLINICAL TRIAL: NCT00342290
Title: Early Pregnancy Evaluation by Three-Dimensional Ultrasound
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998018; OH98-CH-N018
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-06-29

CONDITIONS: First Trimester Bleeding; Pregnancy
Keywords: Pathophysiological Volume Measurement; Power Doppler Ultrasound; Prediction of Adverse Pregnancy Outcome; Subchorionic Hemorrhage

SUMMARY:
Early pregnancy is associated with numerous physiologic alterations - many of which are required to establish normal pregnancy outcome. Three-dimensional ultrasound may provide new opportunities to better characterize some of these early changes. This noninvasive method allows one to arbitrarily scan through a digital ultrasound volume data, visualize organs from different perspectives, and render anatomical features through computer processing. Retrospective measurement of distances and volumes are even possible in the physical absence of the patient.

New information provided by three-dimensional ultrasound may lead to improved understanding about how to counsel parents regarding early pregnancy complications such as bleeding. For example, vaginal bleeding complicates approximately 15-20% of first trimester pregnancies. A common association is subchorionic hemorrhage which is associated with increased risk for miscarriage, preterm delivery, preterm premature rupture of membranes, stillbirth, and placental abruption. Several studies have attempted to characterize subchorionic hemorrhage by conventional two-dimensional ultrasound which is not particularly well-suited for accurate measurement of small irregular hematomas. Consequently, there has been considerable debate about the significance of this finding especially in asymptomatic women who undergo prenatal ultrasound examination for other reasons.

This protocol will attempt to identify prognostic indicators of adverse pregnancy outcome. A maximum of 400 pregnant women up to 20 weeks' gestation with sonographically detected subchorionic hemorrhage will be serially studies to characterize sac volume, placental volume, hematoma volume, and placental blood vessel patterns by 3DUS techniques. These results will be correlated with pregnancy outcome, hormonal markers, and placental pathology. This information is expected to improve our understanding of the natural history of subchorionic bleeding and spontaneous miscarriages as well as prognostic factors influencing pregnancy outcome in both symptomatic and asymptomatic women.

DETAILED DESCRIPTION:
Miscarriage is the most common outcome of pregnancy. Vaginal bleeding complicates up to 25% of all pregnancies, and this clinical sign is associated with an increased risk of spontaneous abortion (also known as miscarriage) and other adverse pregnancy outcomes, such as spontaneous preterm labor, preterm premature rupture of the membranes, pre-eclampsia and intrauterine growth restriction. Despite the importance of vaginal bleeding in clinical obstetrics, there is inadequate understanding about the mechanisms leading to vaginal bleeding, and of tests to predict pregnancy outcome in the majority of cases.

A common finding in patients with first trimester vaginal bleeding is subchorionic hemorrhage, which is associated with an increased risk of miscarriage, preterm delivery, preterm premature rupture of membranes, stillbirth, and placental abruption. Previous attempts to characterize subchorionic hemorrhage have used two-dimensional ultrasound, which is not well-suited for accurate measurement of the volume irregular hematomas. It is not surprising that there has been debate about the significance of subchorionic hemorrhage, especially in asymptomatic women undergoing prenatal ultrasound examination for other reasons in which an intrauterine hematoma is found. Three-dimensional ultrasonography has the potential to improve the characterization of volume and location of intrauterine hematomas. This information may be of value in predicting pregnancy outcome.

The Perinatology Research Branch proposes that first trimester bleeding is one of the great obstetrical syndromes; conditions characterized by a collection of signs and symptoms (in this case vaginal bleeding and cramping), with multiple etiologies. We propose that first trimester bleeding may be the result of a hemostatic disorder of the prenatal endometrium (deciduas), caused by pathologic factors including (1) genetic disorders such as chromosomal abnormalities which often is the result in miscarriage in the first trimester of pregnancy; (2) congenital or acquired hemostatic abnormalities due to thrombophilic mutations; (3) abnormal endocrine processes which may lead to dysregulation of endometrial events required for successful pregnancy; (4) abnormal immunological responses in the maternal/embryo/fetal interface. These abnormalities, which could have clinical significance, cannot be investigated with ultrasound. This protocol describes a comprehensive and systematic study of women who present with bleeding during the first trimester of pregnancy, to improve understanding of the relationship between the location and the size of hematomas (with three-dimensional ultrasounds) and the other factors that may determine the subsequent development of adverse pregnancy outcome.

The Branch will execute this protocol by establishing a first-trimester clinic to study patients who present with this common complication of pregnancy. First trimester bleeding is a common and important complication of pregnancy which has been a neglected area of investigation by private and public agencies. We intend to address what has been an orphan area of clinical research.

ELIGIBILITY:
* INCLUSION CRITERIA:

All pregnant subjects will be recruited under informed consent at Hutzel Hospital. The study population for both arms of this protocol will involve pregnant women between the ages of 15 years-old and older at Hutzel Hospital. The ethnic backgrounds are estimated to involve approximately 60 percent Caucasian and 40 percent African American between both sides.

* Accurate pregnancy dating criteria.
* Estimated gestational age less than or equal to 20 weeks' gestation.
* Visible fetus with normal heart rate and rhythm.

EXCLUSION CRITERIA:

* Poor visualization of the fetus due to technical factors (e.g. obesity).
* Risk factors that increase risk for not keeping serial ultrasound appointments.
* Desire not to have vaginal ultrasound scans.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1998-03-22; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Hutzel Women's Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

REFERENCES:
- [Background] Strobino BA, Pantel-Silverman J. First-trimester vaginal bleeding and the loss of chromosomally normal and abnormal conceptions. Am J Obstet Gynecol. 1987 Nov;157(5):1150-4. doi: 10.1016/s0002-9378(87)80280-6. PMID 3688068
- [Background] Stabile I, Campbell S, Grudzinskas JG. Threatened miscarriage and intrauterine hematomas. Sonographic and biochemical studies. J Ultrasound Med. 1989 Jun;8(6):289-92. doi: 10.7863/jum.1989.8.6.289. PMID 2472492
- [Background] Bloch C, Altchek A, Levy-Ravetch M. Sonography in early pregnancy: the significance of subchorionic hemorrhage. Mt Sinai J Med. 1989 Sep;56(4):290-2. PMID 2677693